CLINICAL TRIAL: NCT04131244
Title: In Vitro Follicle Activation of Dormant Follicles in Patient With Premature Ovarian Failure Under 36 Years Old
Brief Title: In Vitro Follicle Activation in Patient With Premature Ovarian Failure Under 36 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: St. Marianna University School of Medicine (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Sezcan Mumusoglu, Assistant Professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HU0616
Record Dates: First submitted 2018-01-13; First posted 2019-10-18 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Activation of Primordial Follicles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: In vitro activation of primordial follicles by PTEN inhibitor and AKT stimulator — After laparoscopic unilateral oophorectomy, ovarian medulla would be dissected from cortex. After fragmentation of 2 cm square ovarian cortex into smaller pieces they would be incubated PTEN inhibitor and AKT stimulator for 48 hours. Finally we will auto graft these fragments beneath to the fallopian tube peritoneal surface.
  Other Names: Laparoscopic unilateral oophorectomy; Laparoscopic auto grafting of ovarian cortex fragments sub-peritoneally

SUMMARY:
This is a clinical trial that the investigators aim to validate In-vitro Activation (IVA) treatment protocol, which was previously defined by Kazuhiro Kawamura (MD) and Aaron Hsueh (PhD), in Turkish patient with Premature Ovarian Insufficiency (POI) under age 36.

DETAILED DESCRIPTION:
The objectives of the study is as following;

* Validation of the previously defined In-Vitro Activation Protocol approach in Turkish patients under 36 years old with Premature Ovarian Insufficiency (POI).
* Giving an opportunity to young POI patient in Turkey for having genetically own baby.
* Primary outcome measure would be live birth.
* For activation of primordial follicles, phosphatase and tensin homolog (PTEN) inhibitor and protein kinase B (AKT) stimulator will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient with POI
* Short amenorrhea period (1 - 2 years)

Exclusion Criteria:

* Having been treated with chemotherapy and/or radiotherapy;
* Having been diagnosed with advanced stage of endometriosis (endometriomas)
* Having been diagnosed with the chronic diseases such as diabetes, cardiac failure, kidney insufficiency, morbid obesity etc..
* Presence of chromosomal abnormality (Turner, Fragile-X etc.)
* Previous multiple laparotomies
* Menopause >10 years
* Accompanied azoospermia

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Live birth | 2 years
  The primary outcome is live birth, defined as the delivery of a live-born infant at 24 weeks of gestation

SECONDARY OUTCOMES:
Follicle growth rate | 1 year
  Number of ovulation induction cycle achieved to growth follicle
M-II oocyte rate | 1 year
  Number of mature oocyte rate among retrieved oocytes
Day 2-3 good quality embryo rate | 1 year
  Good quality embryo rate of fertilized oocytes (2PN)
Clinical pregnancy rate | 2 years
  A clinical pregnancy is a pregnancy that is confirmed by both high levels of human chorionic gonadotropin (hCG) and ultrasound confirmation of a gestational sac or heartbeat (fetal pole)

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University School of Medicine, Department of Ob/Gyn, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No